CLINICAL TRIAL: NCT05793528
Title: The Effect of Ultrasound Guidance on Radiation Dose and Procedure Time in Lumbar Transforaminal Epidural Injection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-SK-YO-20.03.23
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar
Keywords: Lumbar Transforaminal Epidural Injection; Ultrasound Guided Epidural Injection; Radiation Dose; Procedure Time
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Those who had lumbar radicular pain: Patients with lumbar radicular pain identified by inclusion and exclusion criteria
  Interventions: Procedure: Fluoroscopy Guided Transforaminal Epidural Steroid Injection; Procedure: Ultrasound Guided Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Fluoroscopy Guided Transforaminal Epidural Steroid Injection — The patients are positioned prone. The injection site is cleaned with povidone-iodine 3 times and a sterile drape was applied. Short-acting local anesthesia (3 mL of 2% prilocaine) is applied to the skin and subcutaneous tissue. A 3.5-inch, 22-gauge spinal needle is inserted just below the pedicle. It is advanced into the subpedicular space using the coaxial technique under the intermittent guidance of fluoroscopy. The needle position is confirmed through a lateral view. Using lateral views, the needle is placed at the posterior one-third of the foramen. Using the anteroposterior view, one to 2 mL of the contrast agent (300 mg/50 mL iohexol) is given and the distribution pattern is visualized. Once the epidural distribution of the contrast agent is confirmed without vascular flow, a mixture of 8 mg (two mL) of dexamethasone, 1 mL of physiological saline, and 1 mL (0.5%) of bupivacaine hydrochloride is injected.
Procedure: Ultrasound Guided Transforaminal Epidural Steroid Injection — The patients are positioned prone placed. Following the provision of aseptic conditions, the spinous process of the vertebral midline is visualized using a low-frequency convex ultrasound probe. The lateral edge of the relevant vertebral lamina is visualized by sonographic scanning in the horizontal plane. Local anesthesia is applied to the skin and subcutaneous tissue. A 3.5-inch, 22-gauge spinal needle is advanced to the lateral edge of the relevant vertebral lamina under ultrasound image guidance. Then, anteroposterior imaging is performed with fluoroscopy to confirm needle localization when the lamina margin is reached, and the needle is guided into the foramen under the guidance of fluoroscopy. The contrast agent is given and the distribution pattern is visualized. Once the epidural distribution of the contrast agent is confirmed without vascular flow, a mixture of 2 mL of dexamethasone, 1 mL of physiological saline, and 1 mL (0.5%) of bupivacaine hydrochloride is injected.

SUMMARY:
Low back pain is one of the leading causes of disability, and its social burden and economic cost are quite high. Although there are many causes that can lead to low back pain, radicular pain, which develops mostly secondary to lumbar disc hernias, is one of the most common pathologies. Epidural corticosteroid and local anesthetic injections are an important treatment option in the treatment of lumbar radicular pain that does not respond to conservative methods.

For fluoroscopy-guided epidural injections; transforaminal, interlaminar and caudal approaches may be preferred. It is accepted as the superiority of the transforaminal approach that it allows access to the area of pathology, thus to the anterior epidural area where inflammatory mediators are more concentrated, and that it can spread to the target specifically around the inflamed nerve roots.

In transforaminal epidural injections, the use of ultrasound as the sole imaging tool throughout the entire procedure is still not appropriate, as subbony structures cannot be visualized. However, ultrasound can be integrated at any stage of the process. Thus, the relatively inexpensive cost, portability, and ability to show non-osseous tissues of ultrasonography are utilized, particularly in terms of reducing radiation exposure.

Gofeld et al. claimed that ultrasound-guided transforaminal epidural injection could be performed by targeting the posterior part of the vertebral body. However, in cases where the lamina is wide and covers the posterior of the vertebral body, it may not be possible to sonographically view the vertebral body. In addition, although the intervertebral disc is differentiated from the corpus, loss of fluid content in the elderly can cause acoustic shadowing in the disc. This may result in accidental intra-disc injections. Finally, even if the target point is reached, it is not possible to show intravascular spread at this level ultrasonographically. Therefore, in our opinion, this method is unreliable for transforaminal epidural injections. Another study used ultrasound and fluoroscopy together for transforaminal epidural injections. After imaging the lamina of the relevant vertebral level sonographically, the needle is directed to the lateral edge of the lamina, then fluoroscopic imaging is performed after it passes under the lamina with the loss of resistance technique. However, it should be known that the loss of resistance technique is not a suitable and reliable method in transforaminal injections. In addition, since it is not known how far the lamina has progressed after it has passed under the bone, in other words, imaging guidance is disabled in this part of the process.

In our clinic, we use ultrasonography and fluoroscopy methods in an integrated way (hybrid method) for transforaminal epidural injections. For this purpose, we proceed to fluoroscopic imaging immediately after the spinal needle is advanced to the lateral edge of the lamina at the vertebral level where there is pathology with ultrasound. We think that with this method, we continue to stay in the safe window and reduce the radiation dose and procedure time. Based on this, we determined the aim of this study as the effect of including ultrasonography guidance in transforaminal epidural injections on radiation dose and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-70
* Radicular low back pain
* Failure to respond to conservative treatments
* Pain intensity NRS >3/10
* Lumbar nerve root compression due to disc herniation in lumbar MRI
* Agree to participate in the research

Exclusion Criteria:

* Patients younger than 18 years old and over 70 years old
* Patients describing only localized pain in the lower back without radiating to the lower extremities
* Those with nerve root compression due to reasons other than disc herniation
* Those with spondylolisthesis
* Those with transitional vertebrae
* Pregnancy
* Patients with a body mass index over 30
* Patients with bleeding diathesis
* Having a known psychiatric illness diagnosis
* History of allergy to any of the injection substances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will consist of patients who are planned to receive transforaminal epidural steroid injection or erector spina plane block treatment by the clinician, and who want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in NRS (Numeric Rating Scale) | at first hour
  ≥50% reduction in the NRS scores at first hour relative to the initial NRS scores.
Radiation Dose | at first hour
  Radiation dose during the TFESI
Radiation Time | at first hour
  Radiation time during the TFESI
Procedure Time | at first hour
  Procedure time during the TFESI

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP, Bicket MC, Jamison D, Wilkinson I, Rathmell JP. Epidural steroids: a comprehensive, evidence-based review. Reg Anesth Pain Med. 2013 May-Jun;38(3):175-200. doi: 10.1097/AAP.0b013e31828ea086. PMID 23598728
- [Background] Rivera CE. Lumbar Epidural Steroid Injections. Phys Med Rehabil Clin N Am. 2018 Feb;29(1):73-92. doi: 10.1016/j.pmr.2017.08.007. PMID 29173666
- [Background] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064
- [Background] Patrick N, Emanski E, Knaub MA. Acute and Chronic Low Back Pain. Med Clin North Am. 2016 Jan;100(1):169-81. doi: 10.1016/j.mcna.2015.08.015. PMID 26614726
- [Background] Shim E, Lee JW, Lee E, Ahn JM, Kang Y, Kang HS. Fluoroscopically Guided Epidural Injections of the Cervical and Lumbar Spine. Radiographics. 2017 Mar-Apr;37(2):537-561. doi: 10.1148/rg.2017160043. Epub 2016 Dec 9. PMID 27935769
- [Background] Manchikanti L, Benyamin RM, Falco FJ, Kaye AD, Hirsch JA. Do Epidural Injections Provide Short- and Long-term Relief for Lumbar Disc Herniation? A Systematic Review. Clin Orthop Relat Res. 2015 Jun;473(6):1940-56. doi: 10.1007/s11999-014-3490-4. PMID 24515404
- [Background] Ghahreman A, Ferch R, Bogduk N. The efficacy of transforaminal injection of steroids for the treatment of lumbar radicular pain. Pain Med. 2010 Aug;11(8):1149-68. doi: 10.1111/j.1526-4637.2010.00908.x. PMID 20704666
- [Background] Hong JH, Park EK, Park KB, Park JH, Jung SW. Comparison of clinical efficacy in epidural steroid injections through transforaminal or parasagittal approaches. Korean J Pain. 2017 Jul;30(3):220-228. doi: 10.3344/kjp.2017.30.3.220. Epub 2017 Jun 30. PMID 28757923
- [Background] Gofeld M, Bristow SJ, Chiu SC, McQueen CK, Bollag L. Ultrasound-guided lumbar transforaminal injections: feasibility and validation study. Spine (Phila Pa 1976). 2012 Apr 20;37(9):808-12. doi: 10.1097/BRS.0b013e3182340096. PMID 21912311
- [Background] Yang G, Liu J, Ma L, Cai Z, Meng C, Qi S, Zhou H. Ultrasound-guided Versus Fluoroscopy-controlled Lumbar Transforaminal Epidural Injections: A Prospective Randomized Clinical Trial. Clin J Pain. 2016 Feb;32(2):103-8. doi: 10.1097/AJP.0000000000000237. PMID 25803759
- [Background] Provenzano DA, Narouze S. Sonographically guided lumbar spine procedures. J Ultrasound Med. 2013 Jul;32(7):1109-16. doi: 10.7863/ultra.32.7.1109. No abstract available. PMID 23804333